CLINICAL TRIAL: NCT03023800
Title: A Randomized, Open Label, Single Center Study Comparing the Efficacy of Macular Buckle Versus Vitrectomy + Internal Limiting Membrane Peeling + Gas Tamponade on Macular Schisis and Concurrent Macular Detachment in Eyes With Highly Myopia
Brief Title: Effects of Macular Buckle Versus Vitrectomy on Macular Schisis and Macular Detachment in Highly Myopic Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Lu, Director of Fundus Disease Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013meky013(2)
Record Dates: First submitted 2017-01-16; First posted 2017-01-18 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Retinoschisis; Macular Detachment; High Myopia
MeSH Terms: conditions — Retinoschisis | interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buckle (Experimental): Macular buckling and intraocular gas (C3F8) injection.
  Interventions: Procedure: Macular buckling
- Vitrectomy (Active Comparator): Vitrectomy, internal limiting membrane peeling, and gas tamponade (C3F8).
  Interventions: Procedure: Vitrectomy

INTERVENTIONS:
Procedure: Macular buckling — Surgical procedures of macular buckling, drainage of aqueous fluid (0.1-0.2 ml) through limbal paracentesis, and inject gas ( C3F8 100%, 0.2ml-0.3ml) into vitreous body through pars plana, under systemic anesthesia.
  Arms: Buckle
Procedure: Vitrectomy — Surgical procedures of small gauge vitrectomy, internal limiting membrane peeling, and gas (C3F8, 14%) tamponage, under local or systemic anesthesia
  Arms: Vitrectomy

SUMMARY:
Macular schisis associated with macular detachment is a one of the complications of high myopia. There is controversy in the primary treatment for this situation. This study will compare the effects of macular buckling + gas injection versus vitrectomy + internal limiting membrane peeling + gas tamponade in a cohort of highly myopic eyes with macular retinal detachment associated with macular schisis.

DETAILED DESCRIPTION:
A randomized, open label, single center study comparing the efficacy of macular muckle + gas injection versus internal limiting membrane peeling + gas tamponade on macular schisis associated with macular detachment in eyes with high myopia.

ELIGIBILITY:
Inclusion Criteria:

* axial length ≥ 26.5 mm or refractive error (spherical equivalent) ≥ 8.0 diopter
* macular schisis
* macular retinal detachment
* evidence of posterior staphyloma on clinical examination

Exclusion Criteria:

* severe macular scar
* macular detachment which extended to the peripheral retina (i.e., extension beyond the major vascular arcades in more than one quadrant)
* prominent vitreomacular traction
* a history of vitrectomy or macular buckle
* intraocular active hemorrhage or inflammation
* any media opacity which precluded imaging or clinical evaluation of the macula

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01-30 (Actual); Study Completion 2017-10-12 (Actual)

PRIMARY OUTCOMES:
Retinal re-attachment rate | 3 month

SECONDARY OUTCOMES:
Post-operative best corrected visual acuity | 12 month
Post-operative macular structure on optical coherance tomography | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Lin Lu, MD，PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No